CLINICAL TRIAL: NCT04448379
Title: A Phase Ib,Open Label,Multi-center Study to Assess the Efficacy and Safety of JMT101 Combined With Afatinib (or Osimertinib) in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer With EGFR Exon 20 Insertion Mutations
Brief Title: Efficacy and Safety of JMT101 Combined With Afatinib (or Osimertinib) in Patients With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Collaborators: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JMT101-CSP-001
Record Dates: First submitted 2020-06-16; First posted 2020-06-25 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-07

CONDITIONS: Locally Advanced or Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohort (Experimental): Two dose levels of JMT101 combined with afatinib or osimertinib will be tested according to the "3 + 3" dose-escalation design.
  The dose-limiting toxicity (DLT) will be assessed from the first administration to the end of the first cycle (28 days).
  Interventions: Drug: JMT101
- Dose Expansion Cohort (Experimental): Once the effective dose has been determined, an expansion cohort will be opened to evaluate the efficacy and safety of the selected dose.
  Interventions: Drug: JMT101

INTERVENTIONS:
Drug: JMT101 — IV infusion Q2W for 4 weeks (28-day cycles)
  Other Names: Afatinib or Osimertinib

SUMMARY:
This study is a Phase Ib, open label, multi-center study of to evaluate the safety and efficacy of JMT101 combined with EGFR-TKIs (Afatinib or Osimertinib) in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring EGFR exon 20 insertion mutations.

DETAILED DESCRIPTION:
The objective of the trial is to evaluate the safety and efficacy of JMT101 combined with EGFR-TKIs (afatinib or osimertinib) in patients with locally advanced or metastatic NSCLC with EGFR exon 20 insertion mutations.

This study consists of two parts (Stage I and Stage II). Stage I was a dose escalation study, and Stage II was a dose expansion study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed, locally advanced or metastatic NSCLC, harboring an EGFR exon 20 insertion mutation. ( non-irradiable, non-operable);
* No previous treatment or first-line treatment failed NSCLC;
* At least 1 measurable lesion according to RECIST 1.1;
* ECOG score 0 or 1;

Exclusion Criteria:

* Previously treated with EGFR antibody;
* Symptomatic brain metastasis;
* Interstitial pneumopathy;
* Known hypersensitivity to any ingredient of JMT101, afatinib, osimertinib or their excipients;
* Receiving an investigational product in another clinical study within 4 weeks;
* History of serious systemic diseases;
* History of serious autoimmune diseases;
* Pregnancy or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE V5.0)). | From enrollment until 30 days after the last dose

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Assessed by Blinded Independent Review Committee (IRC) per RECIST Version 1.1 | From first dose to disease progression or end of study, an average of 1 year
Disease control rate (DCR). | From first dose to disease progression or end of study, an average of 1 year
Progression free survival (PFS). | From first dose to disease progression or end of study, an average of 1 year
Overall survival (OS). | From first dose to death or end of study, an average of 1 year
Area under the concentration curve from time 0 to the concentration at last time point (AUC0-last) of JMT101. | From enrollment until 30 days after the last dose
Maximum measured plasma concentration (Cmax) of JMT101. | From enrollment until 30 days after the last dose
Time to maximum plasma concentration (Tmax) of JMT101. | From enrollment until 30 days after the last dose
Half-life (T1/2) of JMT101. | From enrollment until 30 days after the last dose
Immunogenicity profile of JMT101. | From enrollment until 30 days after the last dose
  Blood samples will be collected from subjects post treatment for assessment to detect the presence of anti-drug antibodies and neutralizing antibodies.
Potential biomarkers detected in plasma circulating tumor DNA. | From enrollment up to disease progression, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Chinese Pla General Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing
  - Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Shanghai Chest Hospital, Shanghai Jiaotong University, Shanghai
  - Shanxi Bethune Hospital (Shanxi Academy of Medical Sciences), Taiyuan
  - Shanxi Province Cancer Hospital, Taiyuan
  - Union Hospital, affiliated with TongJi Medical College, HuaZhong University of Science and Technology, Wuhan

REFERENCES:
- [Derived] Zhao S, Zhuang W, Han B, Song Z, Guo W, Luo F, Wu L, Hu Y, Wang H, Dong X, Jiang D, Wang M, Miao L, Wang Q, Zhang J, Fu Z, Huang Y, Xu C, Hu L, Li L, Hu R, Yang Y, Li M, Yang X, Zhang L, Huang Y, Fang W. Phase 1b trial of anti-EGFR antibody JMT101 and Osimertinib in EGFR exon 20 insertion-positive non-small-cell lung cancer. Nat Commun. 2023 Jun 12;14(1):3468. doi: 10.1038/s41467-023-39139-4. PMID 37308490